CLINICAL TRIAL: NCT03966235
Title: Effects of Melatonin on Progression of Coronary Artery Calcification
Brief Title: Melatonin on Coronary Artery Calcification
Acronym: MelonCAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Wei Ren, MD, Prof., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MelonCAC
Record Dates: First submitted 2019-05-26; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Calcification
Keywords: melatonin; coronary artery calcification; adjuvant therapy
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Melatonin group (Experimental): drug: melatonin tablets (Sigma-Aldrich Co. LLC, St. Louis, MO, USA); the frequency:3mg melatonin tablet was taken daily; duration: study treatment was maintained for 6 months.
  Interventions: Drug: Melatonin 3 mg
- Control group (Placebo Comparator): drug: placebo tablet; the frequency: placebo tablet was taken daily; duration: study treatment was maintained for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin 3 mg — Melatonin was taken daily for 6 months.
  Other Names: melatonin
  Arms: Melatonin group
Drug: Placebo — Placebo tablet was taken daily for 6 months.
  Arms: Control group

SUMMARY:
We planned to evaluate the effects of melatonin on progression of coronary artery calcification (CAC) in patients with moderate calcified coronary atherosclerosis.

DETAILED DESCRIPTION:
CAC is prevalent in coronary artery disease (CHD), and the extent of CAC predicts cardiovascular risk. The causes of CAC include dysregulated matrix metabolism, epitaxial mineral deposition, inflammation, oxidative stress, and apoptosis. Melatonin is the main indoleamine produced by the pineal gland; it is known recently to have anti-inflammatory, anti-cancer and antioxidant activities. Several studies have shown that melatonin protects against inflammation and apoptosis in vascular calcification. Melatonin also inhibits oxidative stress-induced apoptosis and calcification in endplate chondrocytes. The investigators planned to determine the efficacy of melatonin on progression of coronary artery calcification (CAC) in patients with moderate calcified coronary atherosclerosis. This study may shed light as to whether oral melatonin supplementation can be an adjunct therapy in CAC patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with a documented Agatston score≥30 and moderate calcified coronary atherosclerosis (<50% diameter lumen narrowing) were eligible for the study.

Exclusion Criteria:

1. unstable angina pectoris
2. symptomatic chronic heart failure and/or left ventricular ejection fraction (EF) <40%
3. atrial fibrillation or other arrhythmias
4. type I diabetes mellitus or uncontrolled type II diabetes mellitus
5. renal failure
6. liver disease
7. gastrointestinal disease that affected absorption

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
a change in CAC score at 6 months measured by coronary CTA | at 6 months
  The primary efficacy endpoint was the effect of melatonin on the change in CAC score at 6 months compared with placebo.

SECONDARY OUTCOMES:
high-sensitivity C-reactive protein (hsCRP) level | at 6 months
  a change in high-sensitivity C-reactive protein (hsCRP) level at 6 months after treatment.
malondialdehyde (MDA) level | at 6 months
  a change in malondialdehyde (MDA) level at 6 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: yu jie zhou, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- PLA general hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilham D, Tsujikawa LM, Sarsons CD, Halliday C, Wasiak S, Stotz SC, Jahagirdar R, Sweeney M, Johansson JO, Wong NCW, Kalantar-Zadeh K, Kulikowski E. Apabetalone downregulates factors and pathways associated with vascular calcification. Atherosclerosis. 2019 Jan;280:75-84. doi: 10.1016/j.atherosclerosis.2018.11.002. Epub 2018 Nov 14. PMID 30476723
- [Background] Shobeiri N, Bendeck MP. Interleukin-1beta Is a Key Biomarker and Mediator of Inflammatory Vascular Calcification. Arterioscler Thromb Vasc Biol. 2017 Feb;37(2):179-180. doi: 10.1161/ATVBAHA.116.308724. No abstract available. PMID 28122774
- [Background] Fernandez A, Ordonez R, Reiter RJ, Gonzalez-Gallego J, Mauriz JL. Melatonin and endoplasmic reticulum stress: relation to autophagy and apoptosis. J Pineal Res. 2015 Oct;59(3):292-307. doi: 10.1111/jpi.12264. Epub 2015 Aug 9. PMID 26201382
- [Background] Dehdashtian E, Mehrzadi S, Yousefi B, Hosseinzadeh A, Reiter RJ, Safa M, Ghaznavi H, Naseripour M. Diabetic retinopathy pathogenesis and the ameliorating effects of melatonin; involvement of autophagy, inflammation and oxidative stress. Life Sci. 2018 Jan 15;193:20-33. doi: 10.1016/j.lfs.2017.12.001. Epub 2017 Dec 5. PMID 29203148
- [Result] Wang Z, Ni L, Wang J, Lu C, Ren M, Han W, Liu C. The protective effect of melatonin on smoke-induced vascular injury in rats and humans: a randomized controlled trial. J Pineal Res. 2016 Mar;60(2):217-27. doi: 10.1111/jpi.12305. Epub 2016 Jan 13. PMID 26681403